CLINICAL TRIAL: NCT05125952
Title: Assessing Ventilator Safety in Patients on Pressure-Support Ventilation
Acronym: ASOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00106860
Record Dates: First submitted 2021-11-08; First posted 2021-11-18 (Actual); Results first posted 2025-10-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-09

CONDITIONS: Acute Respiratory Failure; Mechanical Ventilation Complication; Ventilator-Induced Lung Injury
Keywords: Self-induced lung injury; Pressure-support ventilation
MeSH Terms: conditions — Ventilator-Induced Lung Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Acute Respiratory Failure (Experimental): Patients with acute respiratory failure managed with pressure-support ventilation.
  Interventions: Device: Viasys Avea Ventilator; Device: Philips Respironics NM3 device; Device: Servo U ventilator; Device: Vyaire SmartCath adult nasogastric tube with Esophageal balloon

INTERVENTIONS:
Device: Viasys Avea Ventilator — Measuring dynamic airway driving pressure and static airway driving pressure during pressure support breath, and static airway driving pressure during a volume control breath. Measuring airway occlusion pressure during pressure support breath.
Device: Philips Respironics NM3 device — Measuring static airway driving pressure during pressure support breath
Device: Servo U ventilator — Measuring static airway driving pressure and p0.1 during pressure support breath.
Device: Vyaire SmartCath adult nasogastric tube with Esophageal balloon — Measuring static and dynamic esophageal driving pressure during pressure support breath, and esophogeal pressure change during airway occlusion maneuver.

SUMMARY:
ASOP is a prospective cohort study comparing three methods for assessing risk of self-induced lung injury in patients with acute respiratory failure being managed with pressure-support ventilation. We will describe the relationship between three different assessment methods for risk of self-induced lung injury and compare them to a gold standard measurement.

DETAILED DESCRIPTION:
Ventilator-induced lung injury (VILI) is known to cause significant morbidity and mortality in patients with acute respiratory failure. Most studies on VILI have involved the effects of inappropriate (often excessive) mechanical ventilator settings. More recently, it has been noted that similar lung damage can be caused by large, patient generated, uncontrolled tidal volumes and driving pressures, which has been termed "self-induced lung injury," or SILI.

Pressure-support ventilation (PSV) is a common mechanical ventilation mode often used in patients with active inspiratory efforts to help reduce patient inspiratory work and improve comfort. PSV effectively allows spontaneously breathing patients to determine their breath flow-rate and breath duration, eliminating flow and cycle dyssynchrony. However, pressure support ventilation does not allow for physicians to control tidal volume or driving pressure. The risk of SILI may thus be increased with PSV.

Several different methods have been proposed to address these challenges. However, to date none of these methods have been compared to assess for concordance in their ability to indicate an increased risk of self-induced lung injury. ASOP is a prospective cohort study comparing three methods for assessing risk of self-induced lung injury in patients with acute respiratory failure being managed with pressure-support ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients age ≥18 years with acute respiratory failure receiving invasive mechanical ventilation
* Managed in pressure-support mode of ventilation

Exclusion Criteria:

* Actively undergoing a spontaneously awakening trial or SAT
* Patient or surrogate is unable to provide informed consent
* Currently pregnant
* Currently incarcerated
* Acute exacerbation of an obstructive lung disease
* Known esophageal varices or any other condition for which the attending physician deems an orogastric catheter to be unsafe
* Esophageal, gastric or duodenal surgical procedures within the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-02-08 (Actual); Primary Completion 2023-11-21 (Actual); Study Completion 2023-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil R MacIntyre, MD, Principal Investigator — Professor of Medicine
Locations (1):
- Duke University Hospital, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beitler JR, Malhotra A, Thompson BT. Ventilator-induced Lung Injury. Clin Chest Med. 2016 Dec;37(4):633-646. doi: 10.1016/j.ccm.2016.07.004. Epub 2016 Oct 14. PMID 27842744
- [Background] Slutsky AS, Ranieri VM. Ventilator-induced lung injury. N Engl J Med. 2013 Nov 28;369(22):2126-36. doi: 10.1056/NEJMra1208707. No abstract available. PMID 24283226
- [Background] Sottile PD, Albers D, Smith BJ, Moss MM. Ventilator dyssynchrony - Detection, pathophysiology, and clinical relevance: A Narrative review. Ann Thorac Med. 2020 Oct-Dec;15(4):190-198. doi: 10.4103/atm.ATM_63_20. Epub 2020 Oct 10. PMID 33381233
- [Background] Grieco DL, Menga LS, Eleuteri D, Antonelli M. Patient self-inflicted lung injury: implications for acute hypoxemic respiratory failure and ARDS patients on non-invasive support. Minerva Anestesiol. 2019 Sep;85(9):1014-1023. doi: 10.23736/S0375-9393.19.13418-9. Epub 2019 Mar 12. PMID 30871304
- [Background] Hess DR. Ventilator waveforms and the physiology of pressure support ventilation. Respir Care. 2005 Feb;50(2):166-86; discussion 183-6. PMID 15691390
- [Background] Mauri T, Yoshida T, Bellani G, Goligher EC, Carteaux G, Rittayamai N, Mojoli F, Chiumello D, Piquilloud L, Grasso S, Jubran A, Laghi F, Magder S, Pesenti A, Loring S, Gattinoni L, Talmor D, Blanch L, Amato M, Chen L, Brochard L, Mancebo J; PLeUral pressure working Group (PLUG-Acute Respiratory Failure section of the European Society of Intensive Care Medicine). Esophageal and transpulmonary pressure in the clinical setting: meaning, usefulness and perspectives. Intensive Care Med. 2016 Sep;42(9):1360-73. doi: 10.1007/s00134-016-4400-x. Epub 2016 Jun 22. PMID 27334266

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized to different sequences of receiving the 4 different measurement methods: Viasys Avea Ventilator, Philips Respironics NM3 device, Servo U ventilator, and Vyaire SmartCath adult nasogastric tube with Esophageal balloon.
Period: Overall Study
Arm/Group | Acute Respiratory Failure
Started | 16
Viasys Avea Ventilator | 15
Philips Respironics NM3 Device | 15
Servo U Ventilator | 15
Vyaire SmartCath Adult Nasogastric Tube With Esophageal Balloon | 15
Completed | 15
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: Participants who completed the study.
Arm/Group | Acute Respiratory Failure
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 7
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 63 [37 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 10
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Respiratory System Driving Pressure Measure by Servo Ventilator (DPrs-servo)
Description: Driving pressure in centimeters of water measured with inspiratory hold on Servo Ventilator in pressure-support ventilation.
Time Frame: Study day 1
Measure: Mean (Standard Deviation); unit: centimeters of water
Arm/Group | Acute Respiratory Failure
Number analyzed (Participants) | 15
centimeters of water | 12.3 (2.9)

2. Primary Outcome: Respiratory System Driving Pressure Measure by Respironics NM3 Device (DPrs-NM3)
Description: Driving pressure in centimeters of water measured with Phillips Respironics NM3 device in pressure-support ventilation.
Time Frame: Study day 1
Population: Not measured in 6 patients after Philips announced discontinuation of support for NM3.
Measure: Mean (Standard Deviation); unit: centimeters of water
Arm/Group | Acute Respiratory Failure
Number analyzed (Participants) | 9
centimeters of water | 8.8 (3.2)

3. Primary Outcome: Airway Occlusion Test (AOC)
Description: Maximum negative airway pressure in centimeters of water during an airway occlusion maneuver. The Vyaire SmartCath adult nasogastric tube with esophageal balloon was used to measure esophogeal pressure change during airway occlusion maneuver.
Time Frame: Study day 1
Measure: Mean (Standard Deviation); unit: centimeters of water
Groups:
- Acute Respiratory Failure - Esophageal Balloon: Patients with acute respiratory failure managed with pressure-support ventilation.
  Vyaire SmartCath adult nasogastric tube with Esophageal balloon: Measuring static and dynamic esophageal driving pressure during pressure support breath, and esophogeal pressure change during airway occlusion maneuver.
Arm/Group | Acute Respiratory Failure - Esophageal Balloon
Number analyzed (Participants) | 15
centimeters of water | 17.4 (10.1)

4. Primary Outcome: Respiratory System Driving Pressure Measured During Volume Control Breath.
Description: Airway driving pressure in centimeters of water measured with inspiratory hold in volume control/assist control.
Time Frame: Study day 1
Measure: Mean (Standard Deviation); unit: centimeters of water
Arm/Group | Acute Respiratory Failure
Number analyzed (Participants) | 15
centimeters of water | 12.3 (3.4)

5. Primary Outcome: Transpulmonary Driving Pressure Measured During Volume Control Breath.
Description: Transpulmonary driving pressure in centimeters of water measured via esophageal balloon with inspiratory hold in volume control/assist control.
Time Frame: Study day 1
Population: Not measured in 7 patients who could not have esophageal balloon placed.
Measure: Mean (Standard Deviation); unit: centimeters of water
Arm/Group | Acute Respiratory Failure
Number analyzed (Participants) | 8
centimeters of water | 9.5 (3.6)

6. Secondary Outcome: Duration of Mechanical Ventilation
Description: Number of days receiving mechanical ventilation
Time Frame: Index hospitalization (up to 28 days)
Population: Not measured in 3 patients who were never extubated.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Acute Respiratory Failure
Number analyzed (Participants) | 12
days | 12.4 (9.1)

7. Secondary Outcome: Duration of Intensive Care Unit Admission
Description: Number of days admitted to intensive care unit
Time Frame: Index hospitalization (up to 28 days)
Population: Not measured for 5 patients who did not survive to ICU discharge.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Acute Respiratory Failure
Number analyzed (Participants) | 10
days | 17.2 (6.9)

8. Secondary Outcome: Duration of Hospital Admission
Description: Number of days admitted to hospital
Time Frame: Index hospitalization (up to 28 days)
Population: Not measured in 8 patients who did not survive to hospital discharge.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Acute Respiratory Failure
Number analyzed (Participants) | 7
days | 28 (0.8)

9. Secondary Outcome: Ventilator Free Days
Description: Number of days free from mechanical ventilation
Time Frame: Index hospitalization (up to 28 days)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Acute Respiratory Failure
Number analyzed (Participants) | 15
days | 16 [0 to 21.5]

10. Secondary Outcome: In-hospital Survival
Description: Survival to discharge
Time Frame: Index hospitalization (up to 28 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Acute Respiratory Failure
Number analyzed (Participants) | 15
Participants | 7

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Acute Respiratory Failure
All-Cause Mortality (participants affected / at risk) | 8/15
Serious Adverse Events (participants affected / at risk) | 1/15
Other Adverse Events (participants affected / at risk) | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acute Respiratory Failure (N=15)
Agitation (Nervous system disorders) | 1 (1) — One patient became agitated due to study measurements that required an increase in the dose of sedative medication that they were using.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-05-26): https://cdn.clinicaltrials.gov/large-docs/52/NCT05125952/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-25): https://cdn.clinicaltrials.gov/large-docs/52/NCT05125952/SAP_001.pdf